CLINICAL TRIAL: NCT01376037
Title: An Evaluation of the Effectiveness of the Erchonia ML Scanner (MLS) as a Non-invasive Dermatological Aesthetic Treatment for the Reduction of Circumference of the Upper Arms Clinical Study
Brief Title: Efficacy Study of the Effect of Low Level Laser Light Therapy on Reducing Upper Arm Circumference
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC_ARMBC
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Results first posted 2013-05-29 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Body Contouring
Keywords: upper arm; body contouring; body shaping

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- inactive placebo laser device (Placebo Comparator): The inactive placebo laser device looks identical to the active laser device, but does not emit any therapeutic light output.
  Interventions: Device: inactive placebo laser device
- Erchonia ML Scanner (MLS) (Active Comparator): The Erchonia ML Scanner (MLS) is a low level laser light therapy device comprising 4 independent rotating diodes, each emitting 17mW 635nm of red laser light. The diodes are mounted in scanner devices positioned 120 degrees apart from each other, tilted at a 30 degree angle. The Erchonia® MLS is activated for 20 minutes per arm during which time the 4 rotating diodes create a spiraling circle pattern that is totally random and independent from the others. These patterns overlap each other to guarantee total coverage within the target area. The total laser energy the test subject is exposed to per treated arm is approximately 3.94 joules per square centimeter. Six procedures are administered evenly across 2 weeks.
  Interventions: Device: Erchonia(r) ML Scanner (MLS)

INTERVENTIONS:
Device: Erchonia(r) ML Scanner (MLS) — The Erchonia ML Scanner (MLS) low level laser light therapy device is administered to both arms for 20 minutes each, 6 times across 2 weeks.
  Arms: Erchonia ML Scanner (MLS)
Device: inactive placebo laser device — non-therapeutic light application
  Arms: inactive placebo laser device

SUMMARY:
The purpose of this study is to determine if the Erchonia® ML Scanner (MLS) low level light laser device can help to reduce the circumference of the upper arms.

DETAILED DESCRIPTION:
Upper arm body contouring is designed to remove excess skin and/or fatty tissue from the upper arms. Cosmetic procedures are growing in prevalence, upper arm body contouring procedures increased 4059% from 2000 to 2008, and in 2009, just over 16,100 upper arm lifts were performed in the United States (U.S.). Currently available procedures to reduce upper arm circumference include brachioplasty (arm lift), a surgical procedure to remove excess skin and fatty tissue from the upper arm; liposuction of localized fatty deposits in the upper arm; and diet and exercise to reduce excess body fat. Both brachioplasty and liposuction are surgical procedures with risks and potential complications including trauma; fluid accumulation requiring drainage; injury to the skin; infection; permanent scars; and complications from anesthesia. Low level laser light therapy offers a safe, non-invasive and essentially risk-free alternative to reducing upper arm circumference.

The device being evaluated for the reduction of upper arm circumference, the Erchonia ML Scanner (MLS) is cleared by the Food and Drug Administration (FDA) under K082609 for "... use as a non-invasive dermatological aesthetic treatment for the reduction of circumference of hips, waist, and thighs." Furthermore, FDA identifies this generic type of device as: "A Low Level Laser System for Aesthetic Use is a device using low level laser energy for the disruption of adipocyte cells within the fat layer for the release of fat and lipids from these cells for non-invasive aesthetic use." Therefore, the biochemical effect of the Erchonia® MLS low level laser light therapy device stimulates the mitochondria of the adipocyte cells which in turn increases the production of Adenosine-5'-triphosphate (ATP). The newly synthesized ATP triggers the up-regulation of cyclic adenosine monophosphate (cAMP). cAMP has been shown to stimulate cytoplasmic lipase, triggering the conversion of triglycerides into fatty acids and glycerol that can easily pass through the cell membrane. The transitory pore is evidence that the laser is allowing for the movement of fatty acids, glycerol, and triglycerides to pass across the membrane and into extra-cellular space. Through vasodilation of nearby blood vessels and arteries, oxidization of the triglycerides and fatty acids occurs within the extra-cellular space.

ELIGIBILITY:
Inclusion Criteria:

* Subject indicated for liposuction, or use of liposuction techniques, for the removal of localized deposits of adipose tissues that do not respond to diet and exercise; specifically for the indication of body contouring of the bilateral upper arms (As per the American Academy of Cosmetic Surgery's 2006 Guidelines for Liposuction Surgery developed by A joint Ad Hoc Committee of the American Society of Liposuction Surgery (ASLSS) and the American Academy of Cosmetic Surgery (AACS)), and/or for the procedure of brachioplasty (upper arm lift).
* Body Mass Index (BMI) of 20 to 35 kg/m².
* Subject is willing and able to abstain from partaking in any treatment other than the study procedure to promote body contouring and/or weight loss during study participation.
* Subject is willing and able to maintain his or her regular (typical pre-study procedure) diet and exercise regimen without effecting significant change in either direction during study participation.

Exclusion Criteria:

* Subject is seeking upper arm body contouring as a means of weight loss.
* Diabetes dependent on insulin or oral hypoglycemic medications.
* Known cardiovascular disease such as cardiac arrhythmias, congestive heart failure.
* Cardiac surgeries such as cardiac bypass, heart transplant surgery, pacemakers.
* Prior surgical intervention for body sculpting of the arms, such as liposuction or brachioplasty.
* Prior surgical intervention for weight loss, such as stomach stapling, lap band surgery.
* Medical, physical, or other contraindications for body sculpting/weight loss.
* Current use of medication(s) known to affect weight levels and/or to cause bloating or swelling and for which abstinence during the course of study participation is not safe or medically prudent.
* Any medical condition known to affect weight levels and/or to cause bloating or swelling.
* Mastectomy or operations in the axilla lymph nodes.
* Active infection, wound or other external trauma to the areas to be treated with the laser.
* Pregnant, breast feeding, or planning pregnancy prior to the end of study participation.
* Serious mental health illness such as Alzheimer's, schizophrenia and bipolar disorder; psychiatric hospitalization in past two years.
* Developmental disability or cognitive impairment that in the professional judgment of the study Principal Investigator (PI) would preclude adequate comprehension of the informed consent form and/or ability to record the necessary study measurements.
* Photosensitivity disorder.
* Active or recurrent cancer or currently receiving chemotherapy or radiation therapy.
* Involvement in litigation/worker's compensation claim/receiving disability benefits related to weight-related and/or body shape issues.
* Participation in any type of research in the past 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nestor, M.D.,Ph.D., Principal Investigator; Shari Sanchez, M.D., Principal Investigator — unaffilliated

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty-two (62) subjects were recruited and enrolled between March 21, 2011 and November 28, 2011 at two separate clinical research centers.
Pre-assignment Details: There were no significant events or approaches for the overall study following participant enrollment, but prior to group assignment. There were no enrolled participants excluded from the trial before group assignment and no criteria for this possibility was included in the study design.
Groups:
- Erchonia ML Scanner (MLS): The Erchonia ML Scanner (MLS) is a low level laser light therapy device comprising 4 independent rotating diodes, each emitting 17 milliWatts (mW) 635nm red laser light. The diodes are mounted in scanner devices positioned 120 degrees tileted from each other at a 30 degree angle. The Erchonia® MLS is activated for 20 minutes per arm during which time the 4 rotating diodes create a spiraling circle pattern totally random and independent from the others. These patterns overlap each other to guarantee total coverage within the target area. The total laser energy the test subject is exposed to per treated arm is approximately 3.94 joules per square centimeter.
- Inactive Placebo Laser Device: The inactive placebo laser device looks identical to the active laser device, but does not emit any therapeutic light output.
  inactive placebo laser device : The inactive placebo laser device looks identical to the active laser device, but does not emit any therapeutic light output.
Period: Overall Study
Arm/Group | Erchonia ML Scanner (MLS) | Inactive Placebo Laser Device
Started | 31 | 31
Completed | 31 | 29
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Erchonia ML Scanner (MLS): The Erchonia ML Scanner (MLS) is a low level laser light therapy device comprising 4 independent rotating diodes, each emitting 17mW 635nm ed laser light. The diodes are mounted in scanner devices positioned 120 degrees apart from each other, tilted at a 30 degree angle. The Erchonia® MLS is activated for 20 minutes per arm during which time the 4 rotating diodes create a spiraling circle pattern that is totally random and independent from the others. These patterns overlap each other to guarantee total coverage within the target area. The total laser energy the test subject is exposed to per treated arm is approximately 3.94 joules per square centimeter.
  Erchonia(r) ML Scanner (MLS) : The Erchonia ML Scanner (MLS) is a low level laser light therapy device comprising 4 independent rotating diodes, each emitting 17mW 635nm of red laser light. The diodes are mounted in scanner devices positioned 120 degrees apart from each other, tilted at a 30 degree angle. The Erchonia® MLS is a
- Total: Total of all reporting groups
Arm/Group | Erchonia ML Scanner (MLS) | Inactive Placebo Laser Device | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 31 | 62
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.90 (10.59) | 46.68 (13.11) | 46.29 (11.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 31 | 31 | 62

OUTCOME MEASURES:

1. Primary Outcome: Change in Combined Upper Arm Circumference Measurements From Baseline to Endpoint
Description: Change in combined upper arm circumference measurements is calculated as the difference in combined upper arm circumference measurements from baseline to endpoint (2 weeks) for each of the right upper arm and the left upper arm, separately. A change of at least +1.25 centimeters, for each of the right upper arm and the left upper arm, separately, is considered positive for study success for an individual subject. It was pre-determined that the overall study would be considered a success if at least 50% (16 or more out of 31) of the test group subjects attained individual subject success and individual subject successes in the placebo group were at least 35% lower than for test group subjects (5 or less out of 31).
Time Frame: baseline and 2 weeks
Measure: Number; unit: participants
Arm/Group | Erchonia ML Scanner (MLS) | Inactive Placebo Laser Device
Number analyzed (Participants) | 31 | 31
participants | 18 | 1

ADVERSE EVENTS:
Arm/Group | Erchonia ML Scanner (MLS) | Inactive Placebo Laser Device
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31
Other Adverse Events (participants affected / at risk) | 0/31 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No